CLINICAL TRIAL: NCT00441792
Title: A Randomized Trial of Etomidate Versus Midazolam for Intubation of Patients With Sepsis.
Brief Title: The Effect of Etomidate on Patient Outcomes After Single Bolus Doses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advocate Hospital System (Other)
Collaborators: Emergency Medicine Foundation (Other)
Responsible Party: Principal Investigator, Erik Kulstad, MD, MS, Research Director, Advocate Hospital System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4257
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Results first posted 2012-04-06 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Sepsis; Trauma
Keywords: Sepsis; Etomidate; midazolam; ketamine
MeSH Terms: conditions — Sepsis; Wounds and Injuries | interventions — Etomidate; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Etomidate (Experimental)
  Interventions: Drug: Etomidate
- midazolam (Experimental)
  Interventions: Drug: midazolam

INTERVENTIONS:
Drug: Etomidate — Etomidate at induction dose based on weight
  Arms: Etomidate
Drug: midazolam — Midazolam at induction dose based on weight
  Arms: midazolam

SUMMARY:
The primary aim is to determine the difference in hospital length of stay between septic patients given etomidate and those given midazolam for induction during rapid sequence intubation (RSI) in the emergency department. To achieve this aim we plan to perform a prospective randomized trial measuring the length of stay of patients meeting sepsis criteria and requiring intubation. The investigators will compare in-hospital mortality rates between patients given etomidate and patients given midazolam for induction. In addition to hospital length of stay, secondary endpoints between the two groups will include length of stay in the intensive care unit, death within 48 hours of admission, and total number of days intubated.

Research Hypothesis:

In adult patients presenting to the emergency department with sepsis and requiring rapid sequence intubation, the length of stay of patients given etomidate will be greater than that of patients given the alternative agent midazolam for induction.

DETAILED DESCRIPTION:
Rationale: Although the use of the drug etomidate for continuous sedation in mechanically ventilated patients was found to have detrimental effects on patient mortality shortly after its introduction into clinical practice, etomidate continues to be widely used as an induction agent for endotracheal intubation. Recent data have called into question the safety of using etomidate for even a single bolus in patients at risk of adrenal insufficiency, emphasizing the fact that single bolus doses of etomidate cause measurable adrenal suppression, and consequently may cause an increase in vasopressor requirements and hospital length of stay. Alternative FDA-approved induction agents, such as midazolam, are claimed by many authors to be safer than etomidate; however, no studies have formally compared these agents.

Research Hypothesis: The investigators hypothesize that in critically ill adult patients presenting to the emergency department with sepsis and requiring rapid sequence intubation, the hospital length of stay of patients given etomidate will be increased compared to patients given midazolam for induction.

Specific Aims: The specific aim is to determine the difference in hospital length of stay between septic patients given etomidate and those given midazolam for induction during rapid sequence intubation in the emergency department. The investigators plan to compare the two groups in terms of length of hospital stay, length of ICU stay, and duration of intubation by performing a prospective, randomized, trial of critically ill patients presenting to the emergency department with sepsis requiring intubation. The investigators will also compare the mortality rates in these two groups while controlling for severity of illness and the use of steroids while hospitalized. Significance: If the use of etomidate to induce anesthesia prior to intubation is found to adversely affect the length of stay of septic patients, a reduction in the length of stay in such patients might be achieved by using alternative agents for induction. The current widespread use of an induction agent that may adversely affect the length of stay of septic patients has significant implications for patient management.

ELIGIBILITY:
Inclusion Criteria:

* All critically ill adult patients who present to the emergency department in need of ventilatory support and having a traumatic or suspected infectious etiology for their illness. Specifically, all patients meeting criteria for severe sepsis, septic shock, or the sepsis syndrome by fulfillment of two of the four criteria for the systemic inflammatory response syndrome (temperature greater than 38.3°C or less than 36°C, heart rate greater than 90, respiratory rate greater than 20 or PaCO2 less than 32, white blood cell count greater than 12,000 or less than 4000 or greater than 10% bands).
* All patients presenting in respiratory distress from a presumed pulmonary source of infection and requiring ventilatory support.
* All patients presenting after any traumatic injury and requiring ventilatory support.

Exclusion Criteria:

* An age less than 18
* Pregnancy
* Do-not-resuscitate status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2007-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik B Kulstad, MD, MS, Study Chair — advocate christ medical center
Locations (1):
- Advocate Christ Medical Center, Oak Lawn, Illinois, United States

REFERENCES:
- [Result] Tekwani KL, Watts HF, Sweis RT, Rzechula KH, Kulstad EB. A comparison of the effects of etomidate and midazolam on hospital length of stay in patients with suspected sepsis: a prospective, randomized study. Ann Emerg Med. 2010 Nov;56(5):481-9. doi: 10.1016/j.annemergmed.2010.05.034. Epub 2010 Sep 15. PMID 20828877

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients eligible for this study were enrolled from November 2007 until May 2009. Patients were eligible if they were older than 18 years, were intubated in the ED, and had a suspected infectious cause for their illness.
Groups:
- Midazolam: Patients received either etomidate or midazolam.
- Etomidate: Patients received either etomidate (0.3 mg/kg) or midazolam (0.1 mg/kg) intravenously before rapid sequence intubation in a double-blind fashion. The dose of each medication was chosen according to current physician practice and previous study findings. Identical study vials containing either etomidate or midazolam, in volume-equivalent concentrations, were prepared by our pharmacy department and stored in kits that also contained a variety of commonly used paralytic agents. Kits were labeled with numbers that reflected the assignment generated by a randomization sequence generator and placed in our automated medication dispensing cabinet (Omnicell, Inc., Mountain View, CA). The remainder of the patients' care, both in the ED and in the ICU, was directed according to the treating physician.
Period: Overall Study
Arm/Group | Midazolam | Etomidate
Started | 59 | 63
Completed | 59 | 61 (2 patients lost to follow up in Etomidate arm due to transfer to outside hospital.)
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Midazolam | Etomidate | Total
Number analyzed (Participants) | 59 | 63 | 122
Age, Customized [Median (Inter-Quartile Range); unit: years] | 73 [60 to 80] | 70 [60 to 83] | 72 [60 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 30 | 53
  Male | 36 | 33 | 69

OUTCOME MEASURES:

1. Secondary Outcome: Mortality
Description: In-hospital mortality.
Time Frame: Duration of hospitalization.
Population: All patients entering into the study were analyzed on an intent to treat basis.
Measure: Number (95% Confidence Interval); unit: percentage of patients dying
Groups:
- Midazolam: Patients received midazolam (0.1 mg/kg) intravenously before rapid sequence intubation in a double-blind fashion. The dose of each medication was chosen according to current physician practice and previous study findings. Identical study vials containing either etomidate or midazolam, in volume-equivalent concentrations, were prepared by our pharmacy department and stored in kits that also contained a variety of commonly used paralytic agents. Kits were labeled with numbers that reflected the assignment generated by a randomization sequence generator and placed in our automated medication dispensing cabinet (Omnicell, Inc., Mountain View, CA). The remainder of the patients' care, both in the emergency department and in the intensive care unit, was directed according to the treating physician.
- Etomidate: Patients received etomidate (0.3 mg/kg) intravenously before rapid sequence intubation in a double-blind fashion. The dose of each medication was chosen according to current physician practice and previous study findings. Identical study vials containing either etomidate or midazolam, in volume-equivalent concentrations, were prepared by our pharmacy department and stored in kits that also contained a variety of commonly used paralytic agents. Kits were labeled with numbers that reflected the assignment generated by a randomization sequence generator and placed in our automated medication dispensing cabinet (Omnicell, Inc., Mountain View, CA). The remainder of the patients' care, both in the emergency department and in the intensive care unit, was directed according to the treating physician.
Arm/Group | Midazolam | Etomidate
Number analyzed (Participants) | 59 | 61
percentage of patients dying | 36 [24 to 49] | 43 [30 to 56]

2. Primary Outcome: Length of Stay
Description: The primary outcome of the study was hospital length of stay.
Time Frame: time in days of hospitalization
Population: All patients entering into the study were analyzed on an intent to treat basis.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Midazolam | Etomidate
Number analyzed (Participants) | 59 | 61
days | 9.5 [4.6 to 16] | 7.3 [3.1 to 13]

ADVERSE EVENTS:
Arm/Group | Midazolam | Etomidate
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/61
Other Adverse Events (participants affected / at risk) | 0/59 | 0/61

LIMITATIONS AND CAVEATS:
Because of limitations in the availability of study investigators and pharmacists, we were unable to enroll all potentially eligible patients, raising the possibility that our study sample was not representative of our entire patient population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes